CLINICAL TRIAL: NCT04518514
Title: Telemedical Risk Assessment and Preoperative Evaluation for Anesthesia During the COVID-19 Pandemic
Brief Title: Telemedical Risk Assessment and Preoperative Evaluation (TAPE)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Collaborators: Docs in Clouds Telecare GmbH (Unknown)
Responsible Party: Principal Investigator, Jan Wienhold, cand. Dr. med., RWTH Aachen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-174
Record Dates: First submitted 2020-07-28; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Patients Undergoing Elective Surgery With Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative evaluation and risk assessment via telemedicine (Experimental)
  Interventions: Device: TAPE-Software

INTERVENTIONS:
Device: TAPE-Software — Telemedical Risk Assessment and Preoperative Evaluation prior to anaesthesia via personal computer

SUMMARY:
The purpose of this study is to assess the feasibility, patient satisfaction and time saving of a telemedical risk assessment and preoperative evaluation for anesthesia.

DETAILED DESCRIPTION:
The preanesthesia evaluation and risk assessment is conducted by an anesthesiologist prior to elective surgery. The physician assesses the patient´s medical records and specifies the individual preoperative procedure in order to minimize the perioperative risks. The on-site meeting is often connected with extended travel time and during the COVID-19 pandemic also with an increased infection risk for the patient. This project was initiated to reduce time efforts on patient site and to reduce possible infection risks. The TAPE-software turns every patients home into a remote facility allowing the physician to conduct the preanesthesia evaluation over distance.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* estimated ASA I/II classification based on the American Society of Anesthesiologists (ASA) classification
* elective surgery
* surgery at least 14 days in the future
* patient access to a Windows-10-based personal computer with webcam

Exclusion Criteria:

* language or cognitive barriers (e.g. dementia, laryngectomy...)
* high risk surgeries with need of postoperative ICU stay
* acute infection with required auscultation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility (as defined below) of telemedical risk assessment and preoperative evaluation in anesthesiology as assessed by a questionnaire. | 6 months
  We focus on the feasibility of a telemedical risk assessment and preoperative evaluation in anesthesiology. We defined feasibility in our scenario as:
  * establishment of a video-audio-connection possible
  * complete assessment of the patients medical records possible
  * assessment of the individual perioperative risk possible
  * physician is put into the position to explain planned procedures and related risks
  * digital documentation possible
  * physician is put into the position to answer patient questions
  * physician can acquire all necessary information
  * digital signature on both sides possible
  Those criteria will be assessed by our questionnaires. After preanesthesia evaluation the patient as well as the physician are asked to answer our online questionnaire (two different ones).
Patient acceptance of a telemedical preanesthesia evaluation as assessed by a questionnaire. | 6 months
  After preanesthesia evaluation the patient is asked to answer our online questionnaire. The questionnaire is partly based on a previously published study (Follmann et al., Technical Support by Smart Glasses During a Mass Casualty Incident: A Randomized Controlled Simulation Trial on Technically Assisted Triage and Telemedical App Use in Disaster Medicine, J Med Internet Res 2019;21(1):e11939).
Patient satisfaction with a telemedical preanesthesia evaluation as assessed by a questionnaire. | 6 months
  We aim to investigate patient satisfaction of a telemedical risk assessment and preoperative evaluation in anesthesiology prior to elective surgery. After preanesthesia evaluation the patient is asked to answer our online questionnaire. The questionnaire is partly based on a previously published study (Follmann et al., Technical Support by Smart Glasses During a Mass Casualty Incident: A Randomized Controlled Simulation Trial on Technically Assisted Triage and Telemedical App Use in Disaster Medicine, J Med Internet Res 2019;21(1):e11939).
Time saving for the patient | 6 months
  We quantify time saving on patient site due to the fact that patients do not have to travel to the hospital anymore.
Time saving for the physician | 6 months
  On physician site we investigate possible time saving due to the implementation of the investigator's software.
Adverse events | 6 months
  Number of patients in whom telemedical preanesthesia evaluation lead to adverse events such as postponed surgery and adverse events during surgery which are caused by the preanesthesia evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Follmann, Dr., Principal Investigator — RWTH Aachen University Hospital; Jan Wienhold, cand. med., Principal Investigator — RWTH Aachen University Hospital
Locations (1):
- RWTH Aachen University Hospital, Aachen, Germany

REFERENCES:
- [Derived] Wienhold J, Mosch L, Rossaint R, Kemper I, Derwall M, Czaplik M, Follmann A. Teleconsultation for preoperative evaluation during the coronavirus disease 2019 pandemic: A technical and medical feasibility study. Eur J Anaesthesiol. 2021 Dec 1;38(12):1284-1292. doi: 10.1097/EJA.0000000000001616. PMID 34669644